CLINICAL TRIAL: NCT07209956
Title: Evaluation de la Valeur Pronostique du TAPSE (Tricuspid Plane Annular Systolic Excursion) Dans la Bronchiolite aigüe sévère Chez l'Enfant hospitalisé en réanimation ou Soins Continus pédiatriques
Brief Title: Etude PROTECT : Prognostic Role of Tapse Evaluation in Children's bronchioliTis
Acronym: PROTECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2022/17
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Bronchiolitis; Viral
Keywords: acute bronchiolitis; echocardiography; TAPSE; myocardial dysfunction; pulmonary hypertension; PICU
MeSH Terms: conditions — Bronchiolitis; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAPSE marker (Experimental): At every admission in PICU for acute bronchiolitis, a screening for inclusion and exclusion factors will be carried out by an investigator. If the patient is included in the study, an echocardiographic assessment with measurement of the TAPSE will be performed, within the 36h following admission. The patient will then be followed until discharge of hospital, or death, or the end of the inclusion period. We will study the association between the TAPSE value at admission, and the PICU length of stay, in order to determine its prognostic role in severe acute bronchiolitis.
  If, during the follow-up period, intubation for invasive ventilation is required, a second echocardiographic assessment will be performed, and the second TAPSE value will be compared to the first one, for exploratory purposes on cardiopulmonary interactions.
  Interventions: Procedure: Echocardiographic assessment of TAPSE

INTERVENTIONS:
Procedure: Echocardiographic assessment of TAPSE — Non interventional study (study of a prognostic factor). The study procedure is the echocardiographic assessment of TAPSE at every admission in PICU for acute bronchiolitis.
  Transthoracic echocardiography is a non invasive, non radiative examination, that is usually performed at every admission in PICU, however not mandatory. Inclusion in the study will lead to a systematic echocardiographic assessment at admission, potentially adding this examination to the patient's course.
  As transthoracic echocardiography is systematically monitored in intubated children, no additional examination will be necessary for those requiring invasive mechanical ventilation.

SUMMARY:
In this prospective study, we aim to evaluate the association between an echocardiographic marker of right ventricular systolic function, the TAPSE (Tricuspid Annular Plane Systolic Excursion), and poor outcome in patients admitted to Pediatric Intensive Care Unit (PICU) for Acute Bronchiolitis (AB).

DETAILED DESCRIPTION:
During the winter season, acute bronchiolitis is the leading cause of PICU admissions among children under the age of 2 years old, worldwide. Indeed, it is estimated that 10% of children hospitalized for AB will require intensive care, with lengths of stay ranging from several days to several weeks. It is therefore crucial to identify those patients at highest risk of severe disease in order to provide the best management options and potentially decrease morbidity. Recently, the prognostic value of the TAPSE (Tricuspid Annular Plane Systolic Excursion), a marker of right ventricle systolic dysfunction, has been demonstrated in adults suffering from SARS-Cov-2 pneumoniae. Indeed, several studies identify a decrease in TAPSE as a marker associated with an increased mortality among patients hospitalized in ICU with SARS Cov-2 pneumoniae. Moreover, some pediatric studies suggest that pulmonary pressures and right ventricular function could be impaired in AB, and thus associated with a less favorable outcome. None of these studies has specifically investigated the TAPSE as a predictor of severity in AB. To address this question, we plan to conduct a prospective study among children admitted to PICU with AB, and evaluate the association between the TAPSE value at PICU admission, and the PICU length of stay. Patients included in the study, will undergo a systematic echocardiographic assessment with measurement of the TAPSE, within the first 36 hours of admission in PICU for AB. They will then be followed until discharge of hospital, or the occurrence of death, or until the end of the inclusion period. If, during the follow-up period, intubation for invasive ventilation is required, a second echocardiographic assessment will be performed, with measurement of the TAPSE, in order to compare it to the initial value, in secondary analysis for exploratory purposes.

ELIGIBILITY:
Inclusion Criteria:

* Infants under the age of 2
* Admitted to PICU with diagnosis of acute bronchiolitis (according to AAP criteria)
* Within the first 36h of PICU stay

Exclusion Criteria:

* Patients suffering from Chronic Heart Disease, chronic respiratory disease (including bronchopulmonary dysplasia and excluding asthma)
* Impairment of echocardiographic window

Ages: 0 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
PICU lenght of stay | Upon discharge from intensive care, maximum of 5 months
  The primary outcome will be the PICU length of stay (LOS), in days.

SECONDARY OUTCOMES:
Hospital length of stay (days) | discharge from the hospital, or until his or her death, maximmum of 5 months
  Hospital length of stay (days)
Intubation and ventilation | Upon discharge from intensive care, maximum of 5 months
  Need for intubation and invasive ventilation during the PICU stay
Respiratory support | Upon discharge from intensive care, maximum of 5 months
  Length of respiratory support (days)
Death | until his or her death, maximum of 5 months
  Patient death

CONTACTS AND LOCATIONS:
Locations (1):
- Bordeaux Hospital University, Bordeaux, France